CLINICAL TRIAL: NCT06820632
Title: From Classrooms to Playgrounds in Bhutan: Evaluating the Role of School-based Physical Education on Physical Fitness, Socio-emotional Competencies and Well-being in Young Adolescents
Brief Title: School-based Physical Education in Bhutan for Physical Fitness and Socio-emotional Competencies in Adolescents
Acronym: ActiveClass-BH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Paro College of Education (Unknown); Royal Thimphu College (Unknown)
Responsible Party: Principal Investigator, Vanessa Siffredi, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CIRSport2025
Record Dates: First submitted 2025-01-29; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: School-based Intervention
Keywords: physical education; adolescence; socio-emotional competencies; well-being; bhutan

STUDY DESIGN:
Intervention Model Description: Two public urban schools will be randomly assigned to either the "enhanced physical education program" or "standard curriculum" condition. An additional "control school", with no physical education, will be included in the study but not in the randomisation process for feasibility concern.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Enhanced physical education (Experimental): The "Enhanced physical education" arm is based on the Health and Physical Education Curriculum Framework developed by the Bhutanese Ministry of Education and well-document in the 2022 edition, www.education.gov.bt. The enhanced PE group will receive two 90-minute sessions weekly for 5 months. The enhanced PE program incorporate both PE with socio-emotional competencies, such as self-regulation, self- and social-awareness, empathy-building exercises, and cooperation activities.
  Interventions: Behavioral: Enhanced physical education
- Health and Physical Education (HPE) standard curriculum (Active Comparator): Health and Physical Education (HPE) standard curriculum is mainly a physical education class limited to a single weekly hour and is highly dependent on the motivation of individual teachers and schools.
  Interventions: Behavioral: HPE Standard curriculum
- Control school (No Intervention): A school without physical education classes

INTERVENTIONS:
Behavioral: Enhanced physical education — The "Enhanced physical education" is based on the Health and Physical Education (HPE) Curriculum Framework developed by the Bhutanese Ministry of Education and well-document in the 2022 edition, www.education.gov.bt. The enhanced PE group will follow closely the description of the HPE curriculum and receive two 90-minute sessions weekly for 5 months. According to the HEP curriculum, the enhanced PE program incorporate both PE with socio-emotional competencies, such as self-regulation, self- and social-awareness, empathy-building exercises, and cooperation activities.
  Arms: Enhanced physical education
Behavioral: HPE Standard curriculum — Health and physical education (HPE) standard curriculum includes roughly one hour per week of general physical education, typically involving activities like football and basketball.
  Arms: Health and Physical Education (HPE) standard curriculum

SUMMARY:
Despite global evidence supporting the benefits of PE in promoting socio-emotional skills, much of the research has focused on countries where PE is a mandatory part of the curriculum. In contrast, Bhutan's Health and Physical Education (HPE) program is limited, with many schools lacking a structured curriculum and dedicated PE educators. This project aims to evaluate the impact of an enhanced school-based physical education (PE) program on physical fitness, socio-emotional competencies, and well-being among upper primary school students in Bhutan.

This project is a methodological collaboration between the Centre Hospitalier Universitaire Vaudois in Switzerland and the Paro College of Education and Royal Thimphu College in Bhutan.

Two public urban schools will be randomly assigned to either the "enhanced physical education program" or "standard curriculum" condition. An additional "control school", with no physical education, will be included in the study but not in the randomisation process for feasibility concern. A total of 360 young adolescents (120 per school, aged 12-14) will be enrolled. Baseline data on individual characteristics such as age, gender, and socio-economic status will be collected through self- and parent-reported questionnaires. Primary outcome measures include physical fitness assessed by PE teachers using various metrics, as well as socio-emotional competencies and well-being evaluated through standardised self- and parent-reported questionnaires. Data will be analysed using an intention-to-treat approach.

This project offers a unique opportunity to explore the international impact of PE within Bhutan's socio-cultural context.

DETAILED DESCRIPTION:
Evidence shows that physical activity, including school-based physical education (PE), supports children's socio-emotional competencies and well-being, including enhancing self-regulation and reducing anxiety and depression. These positive outcomes often vary based on individual factors, including gender and socio-economic status. Given the amount of time children spend in school, this setting provides an ideal platform for enhancing their socio-emotional competencies and well-being through diverse PE opportunities. To date, most research on the association between PE and socio-emotional competencies has been conducted in countries where PE is a mandatory component of the school curriculum, such as those in Europe, the United States, and Australia. Bhutan, a Himalayan Buddhist country with a rich cultural heritage, has seen rapid social changes over the past 20-30 years. Rapid modernisation has led to lifestyle changes among youth, contributing to increasing social issues, sedentary habits and mental health challenges. School-based PE, known as Health and Physical Education (HPE), is limited to a single weekly hour and is highly dependent on the motivation of individual teachers and schools. Anecdotal evidence suggests that many schools do not have a dedicated time slot for HPE. HPE also faces obstacles, including the absence of a structured curriculum, limited trained PE educators, and a lack of prioritisation compared to other subjects.

This project aims to evaluate the impact of a school-based enhanced PE program on physical fitness, socio-emotional competencies and well-being in upper primary school students in Bhutan, compared to a school with HPE standard curriculum and a school with no PE.

This project is a methodological collaboration between the Centre Hospitalier Universitaire Vaudois in Switzerland (Dr Vanessa Siffredi, Dr Russia Hà-Vinh Leuchter) and the Paro College of Education and Royal Thimphu College in Bhutan (Prof. Kezang Sherab and Dr Pema Chopel). The Bhutanese team will implement the intervention and oversee on-site data collection, with the Swiss team providing methodological and statistical support.

Using a randomised controlled trial design, we will assign two urban public schools to either an "enhanced PE", grounded in Bhutan's health and physical education curriculum, or a "HPE standard curriculum" group. An additional "control school", without PE classes, will be included outside of the randomisation for feasibility concern. The study anticipates enrolling n=120 young adolescents per school (total n=360, ages 12- to 14-year-old). The enhanced PE group will receive two 90-minute sessions weekly for 5 months. The enhanced PE program incorporate both PE with socio-emotional competencies, such as self-regulation, self- and social-awareness, empathy-building exercises, and cooperation activities. Baseline individual characteristics (e.g., age, gender, socio-economic status, frequency of physical activity) will be collected pre-intervention via self- and parent-reported questionnaires. Primary outcomes, including physical fitness, socio-emotional skills, well-being, will be measured pre- and post-intervention. Physical fitness will be assessed by PE teachers (muscular strength, muscular endurance, flexibility, cardiorespiratory endurance, balance, coordination, agility, speed and power). Socio-emotional competencies and well-being will be evaluated in the young adolescents using standardised self- and parent-reported questionnaires.

This project offers a unique opportunity to evaluate the international impacts of PE on adolescents' socio-emotional competencies and well-being, especially within Bhutan's distinctive socio-cultural context. Given PE's low prioritisation, findings from this study will be valuable for guiding the Bhutanese national sport curriculum. More broadly, i will contribute to global research on PE and its role in fostering socio-emotional competencies and well-being in youth.

ELIGIBILITY:
Inclusion Criteria:

* Enrolment in participating schools: Students must be enrolled in upper primary school classes (grades 7 and 8) in one of the three participating school.
* Regular school attendance: Students must attend school regularly to ensure consistent exposure to the intervention (min 80% of the courses).
* Parental consent: Written informed consent from a parent or guardian.
* Verbal assent from the child, indicating their willingness to participate.

Exclusion Criteria:

* Inability to participate in physical education courses: Students unable to participate in physical education classes due to medical or other significant reasons.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Socio-emotional competencies: Self-reported, Strength and Difficulty Questionnaire (SDQ) | Pre-intervention (baseline) and 16 weeks post-intervention
  Socio-emotional competencies will be evaluated in young adolescents using the standardised self-reported Strength and Difficulty Questionnaire (SDQ).
  The SDQ is a well-validated 25-item questionnaire designed to assess behavioural problems in children and adolescents aged 4 to 16. It consists of: a) four subscales, emotional symptoms, conduct problems, hyperactivity/inattention, and peer problems (min=0, max=10) with higher scores indicate more difficulties, b) an additional prosocial behavior subscale with higher scores indicate better outcomes in prosocial behavior, and c) a total difficulties score, based on emotional symptoms, conduct problems, hyperactivity/inattention, and peer problems, is also measured with higher scores reflecting greater behavioral difficulties (min=0, max=40).
Socio-emotional competencies: Self-reported, Self-Compassion Scale | Pre-intervention (baseline) and 16 weeks post-intervention
  Socio-emotional competencies will be evaluated in young adolescents using the standardised self-reported Self-Compassion Scale.
  This 26-item scale measures self-compassion across six key dimensions: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. Each item is rated on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). The total score ranges from 26 to 130, with higher scores indicating greater self-compassion and emotional resilience.
Socio-emotional competencies: Self-reported, Empathy Questionnaire for children and adolescents | Pre-intervention (baseline) and 16 weeks post-intervention
  Socio-emotional competencies will be evaluated in young adolescents using the standardised self-reported Empathy Questionnaire for children and adolescents.
  This 15-item scale assesses empathy in adolescents across five dimensions: emotional contagion, self-awareness, perspective-taking, emotional regulation, and empathic action. Each item is scored on a 4-point Likert scale, resulting in a total score ranging from 15 to 60 with higher scores indicate stronger empathy abilities.
Socio-emotional competencies: Self-reported, Self-Efficacy Questionnaire for Youth | Pre-intervention (baseline) and 16 weeks post-intervention
  Socio-emotional competencies will be evaluated in young adolescents using the standardised self-reported Self-Efficacy Questionnaire for Youth.
  This brief questionnaire is designed to assess self-efficacy in youths. It consists of 10 items, each rated on a 5-point Likert scale. The Self-Efficacy Questionnaire for Youth gives a total score that range from 10 to 50, with higher scores reflecting better perceived self-efficacy.
Socio-emotional competencies: Parent-reported, Strength and Difficulty Questionnaire (SDQ) | Pre-intervention (baseline) and 16 weeks post-intervention
  Socio-emotional competencies will be evaluated in young adolescents using the standardised parent-reported Strength and Difficulty Questionnaire (SDQ). The SDQ is a well-validated 25-item questionnaire designed to assess behavioural problems in children and adolescents aged 4 to 16. It consists of: a) four subscales, emotional symptoms, conduct problems, hyperactivity/inattention, and peer problems (min=0, max=10) with higher scores indicate more difficulties, b) an additional prosocial behavior subscale with higher scores indicate better outcomes in prosocial behavior, and c) a total difficulties score, based on emotional symptoms, conduct problems, hyperactivity/inattention, and peer problems, is also measured with higher scores reflecting greater behavioral difficulties (min=0, max=40).
Socio-emotional competencies: Parent-reported, Behaviour Rating Inventory of Executive Function (BRIEF) | Pre-intervention (baseline) and 16 weeks post-intervention
  Socio-emotional competencies will be evaluated in young adolescents using the standardised parent-reported Behaviour Rating Inventory of Executive Function (BRIEF), Behavioural Regulation Scale.
  The Behavioural Regulation Scale from the BRIEF consists of 16 items designed to evaluate a child's ability to control their behaviour and emotions, such as impulse control, emotional regulation, and the capacity to shift between tasks or thoughts.
  The Behavioural Regulation Scale is typically reported as T-scores (M=50, SD=10) with higher scores reflect more executive difficulties.
Socio-emotional competencies: Parent-reported, Social Skills Improvement System (SSIS) | Pre-intervention (baseline) and 16 weeks post-intervention
  Socio-emotional competencies will be evaluated in young adolescents using the standardised parent-reported Social Skills Improvement System (SSIS), Social Skills Scale. The Social Skills Scale from the SSIS consists of 46 items, each rated to reflect the frequency and quality of specific social behaviours in different contexts. It is designed to assess a range of social behaviours that contribute to positive interactions and relationships. This scale evaluates various domains, including communication, cooperation, assertion, responsibility, empathy, engagement, and self-control.
  The instrument yields norm-referenced scores for the Social Skills Scale (M = 100, SD = 15) with higher scores reflecting better social competence and more positive social interactions.
Well-being: Self-reported, KIDSCREEN-27 | Pre-intervention (baseline) and 16 weeks post-intervention
  Well-being will be evaluated in young adolescents using the standardised self-reported KIDSCREEN-27 questionnaire.
  The KIDSCREEN-27 contains 27 items, with responses capturing the frequency or intensity of experiences related to the child's health and well-being over the past week. It is designed to measure health-related quality of life and it assesses five dimensions: Physical Well-being, Psychological Well-being, Autonomy & Parent Relations, Social Support & Peers, and School Environment. For each dimension, scores are typically transformed to a continuous scale ranging from 0 to 100, with higher scores reflecting better outcomes.
Well-being: Parent-reported, KIDSCREEN-27 | Pre-intervention (baseline) and 16 weeks post-intervention
  Well-being will be evaluated in young adolescents using the standardised parent-reported KIDSCREEN-27 questionnaire.
  The KIDSCREEN-27 contains 27 items, with responses capturing the frequency or intensity of experiences related to the child's health and well-being over the past week. It is designed to measure health-related quality of life and it assesses five dimensions: Physical Well-being, Psychological Well-being, Autonomy & Parent Relations, Social Support & Peers, and School Environment. For each dimension, scores are typically transformed to a continuous scale ranging from 0 to 100, with higher scores reflecting better outcomes.
Push-up measurement | Pre-intervention (baseline) and 16 weeks post-intervention
  Push-up (total number of repetitions) will be assessed by PE teachers. This measurement is part of the general physical fitness assessment.
Sit-Up/Curl-Up test | Pre-intervention (baseline) and 16 weeks post-intervention
  Sit-Up/Curl-Up Test (total number of repetitions) will be assessed by PE teachers. This measurement is part of the general physical fitness assessment.
Sit and Reach test | Pre-intervention (baseline) and 16 weeks post-intervention
  Sit and Reach Test (in cm) will be assessed by PE teachers. This measurement is part of the general physical fitness assessment.
Run in Place test | Pre-intervention (baseline) and 16 weeks post-intervention
  Run in Place for 90 seconds (record number of heart rate in 30 seconds) will be assessed by PE teachers. This measurement is part of the general physical fitness assessment.
One foot balance test | Pre-intervention (baseline) and 16 weeks post-intervention
  One foot balance (in seconds) will be assessed by PE teachers. This measurement is part of the general physical fitness assessment.
Basic paper ball bounce test | Pre-intervention (baseline) and 16 weeks post-intervention
  Basic paper ball bounce test (bounce the ball at least three times with each hand) will be assessed by PE teachers. This measurement is part of the general physical fitness assessment.
Left-right paper ball bounce test | Pre-intervention (baseline) and 16 weeks post-intervention
  Bounce the ball back and forth between the right and left hands (maximum number of bouncing) will be assessed by PE teachers. This measurement is part of the general physical fitness assessment.
Shuttle Run test | Pre-intervention (baseline) and 16 weeks post-intervention
  Shuttle Run test (9 meters side move repetitions - number of times/repetitions) will be assessed by PE teachers. This measurement is part of the general physical fitness assessment.
Dash test | Pre-intervention (baseline) and 16 weeks post-intervention
  50 meters Dash test (in seconds) will be assessed by PE teachers. This measurement is part of the general physical fitness assessment.
Standing Broad Jump test | Pre-intervention (baseline) and 16 weeks post-intervention
  Standing Broad Jump (in cm) will be assessed by PE teachers. This measurement is part of the general physical fitness assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Kezang Sherab, PhD, Principal Investigator — Paro College of Education & Royal Thimphu College, Bhutan; Vanessa Siffredi, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV), Switzerland
Locations (1):
- Paro College of Education, Bhutan, Paro, Paro Dzongkhag, Bhutan

IPD SHARING:
Plan to Share IPD: No
Data will be available to researchers who provide a proposal that supports the aims of the approved study. Proposals should be submitted to kezangsherab.pce@rub.edu.bt

REFERENCES:
- [Background] Spruit A, Assink M, van Vugt E, van der Put C, Stams GJ. The effects of physical activity interventions on psychosocial outcomes in adolescents: A meta-analytic review. Clin Psychol Rev. 2016 Apr;45:56-71. doi: 10.1016/j.cpr.2016.03.006. Epub 2016 Apr 3. PMID 27064552
- [Background] Choden U, Sherab K, Howard J. Experience of bullying among Bhutanese college students: implications for teacher formation programmes. Int J Adolesc Med Health. 2019 Nov 25;34(1). doi: 10.1515/ijamh-2019-0087. PMID 31760378
- [Background] Lubans D, Richards J, Hillman C, Faulkner G, Beauchamp M, Nilsson M, Kelly P, Smith J, Raine L, Biddle S. Physical Activity for Cognitive and Mental Health in Youth: A Systematic Review of Mechanisms. Pediatrics. 2016 Sep;138(3):e20161642. doi: 10.1542/peds.2016-1642. Epub 2016 Aug 19. PMID 27542849